CLINICAL TRIAL: NCT01280604
Title: Effects of Fenofibrate 160mg to 54mg Conversion on Triglyceride Levels in Patients on Statin Therapy
Brief Title: Effect of Fenofibrate Conversion on Triglyceride Levels in Patients on Statin Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPGA-10KMani-01
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention 'Fenofibrate 54mg' (Experimental): Subjects in the dose reduction group will be converted from 160mg of fenofibrate to 54mg of fenofibrate daily for 6-8 weeks.
  Interventions: Drug: Fenofibrate 54mg
- Control 'Fenofibrate 160mg' (No Intervention): Subjects in the control group will be remain on 160mg of fenofibrate daily for the duration of the study (6-8 weeks).

INTERVENTIONS:
Drug: Fenofibrate 54mg — Subjects will receive fenofibrate 54mg daily.
  Arms: Intervention 'Fenofibrate 54mg'

SUMMARY:
The primary objective of this randomized trial is to measure the impact of converting patients on statin therapy from fenofibrate 160mg to 54mg per day compared to patients who continue fenofibrate 160mg per day for triglycerides.

DETAILED DESCRIPTION:
Hypothesis: Study subjects receiving fenofibrate 54mg will maintain similar triglyceride levels as patients on 160mg of fenofibrate.

The primary objective of this randomized trial is to measure the impact of converting patients on statin therapy from fenofibrate 160mg to 54mg per day compared to patients who continue fenofibrate 160mg per day for triglycerides. Secondary objectives include evaluating effect of the dosage change on low-density lipoprotein (LDL), HDL, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and serum creatinine (SCr), and the potential cost savings associated with prescribing 54mg instead of 160mg. Electronic medical records will be used to identify subjects and gather data on demographics, comorbid conditions, and concomitant lipid lowering therapy. Subjects will be recruited for enrollment via telephone by the principal investigator (PI), co-principal investigators (Co-PIs), or provider referral after eligibility screening and approval from their primary care physician. Subjects must provide written informed consent and Health Insurance Privacy and Accountability Act (HIPAA) privacy rule authorization prior to participation in this study. Subjects will be randomized to either the intervention arm (conversion to 54mg of fenofibrate) or to the control arm (remain on 160mg of fenofibrate). Subjects in both study arms will have fasting lipid panels, ALT/AST, and SCr evaluated at baseline. All subjects will have repeat labs approximately 8 weeks after enrollment. All subjects will continue to receive standard care based on lipid values. The study period will begin approximately October 29, 2010 and run to June 30, 2011.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Patients actively taking fenofibrate 160mg and statin therapy
* A fasting lipid panel within the past 9 months with most recent triglycerides levels less than 200mg/dL
* Primary care physician approves participation and fenofibrate conversion

Exclusion Criteria:

* Impaired renal function defined as creatine clearance ≤ 50ml/min
* Current enrollment in other studies or clinical trials
* Previous fenofibrate 54mg use
* A history of pancreatitis or known previous triglyceride levels >1000mg/dL
* Pregnancy
* Members with plan benefits that include a deductible for lab services at Kaiser Permanente

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Manigault, PharmD, Principal Investigator — Pharmacy Resident
Locations (1):
- Kaiser Permanente of Georgia, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Subjects in the dose reduction group will be converted from 160mg of fenofibrate to 54mg of fenofibrate daily for 6-8 weeks.
  Fenofibrate 54mg: Subjects will receive fenofibrate 54mg daily.
- Control: Subjects in the control group will be remain on 160mg of fenofibrate daily for the duration of the study (6-8 weeks).
Period: Overall Study
Arm/Group | Intervention | Control
Started | 33 | 33
Subjects Meeting All Inclusion Criteria | 25 | 29
Completed | 24 | 28
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.67) | 57.55 (9.26) | 57.41 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 17 | 22 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 25 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Triglyceride Levels
Description: Triglyceride levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
milligram/deciliter
  Baseline Triglyceride Levels | 135.5 (36.22) | 108.3 (37.41)
  Follow-Up Triglyceride Levels | 152.7 (42.61) | 109 (39.70)

2. Secondary Outcome: Low-density Lipoprotein (LDL)
Description: LDL levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
milligram/deciliter
  Baseline Low-density lipoprotein | 95.32 (21.32) | 83.29 (22.99)
  Follow-up Low-density lipoprotein | 84.42 (21.05) | 78.71 (21.93)

3. Secondary Outcome: High-density Lipoprotein,(HDL)
Description: HDL levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
milligram/deciliter
  Baseline High-density lipoprotein | 41.88 (9.58) | 41.79 (14.24)
  Follow-up High-density lipoprotein | 43.21 (38.99) | 38.79 (33.61)

4. Secondary Outcome: Alanine Aminotransferase(ALT)
Description: ALT levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: international units/liter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
international units/liter
  Baseline Alanine aminotransferase | 29.76 (26.20) | 30.66 (26.61)
  Follow-up Alanine aminotransferase | 27.38 (9.13) | 29.96 (11.03)

5. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: AST levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: international units/liter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
international units/liter
  Baseline Aspartate Aminotransferase | 27.48 (6.14) | 27.59 (8.57)
  Follow-up Aspartate Aminotransferase | 25.5 (5.41) | 26.36 (6.49)

6. Secondary Outcome: Serum Creatinine(SCr)
Description: SCr levels will be assessed in study participants 6-10 weeks after entry into study.
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
milligram/deciliter
  Baseline Serum Creatinine | 0.9880 (0.2571) | 1.14 (0.24)
  Follow-up Serum Creatinine | 1 (0.23) | 1.13 (0.23)

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/29
Other Adverse Events (participants affected / at risk) | 0/25 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No